CLINICAL TRIAL: NCT04481360
Title: Evaluation of Clinical Characteristics and Outcome of COVID19 Pneumonia in Assiut
Brief Title: Evaluation of Clinical Characteristics and Outcome of COVID19 Pneumonia in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Omil Saman, Principle investigator, Assiut University
Other Study IDs: Presentation of COVID19 in AUH
Record Dates: First submitted 2020-07-11; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with covid 19 pneumonia: clinical presentation & outcome of covid 19 pneumonia
  Interventions: Device: CT of the chest

INTERVENTIONS:
Device: CT of the chest — Degree of affection on the lung infected by COVID19

SUMMARY:
* Evaluation of the clinical presentation of COVID 19 pneumonia.
* Identification the risk factors of severing COVID 19 pneumonia.
* Evaluation of the outcome of the disease.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is defined as illness caused by a novel coronavirus now called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; formerly called 2019-nCoV), which was first identified amid an outbreak of respiratory illness cases in Wuhan City, Hubei Province, China. It was initially reported to the WHO on December 31, 2019. On January 30, 2020, the WHO declared the COVID-19 outbreak a global health emergency.On March 11, 2020, the WHO declared COVID-19 a global pandemic, its first such designation since declaring H1N1 influenza a pandemic in 2009. The incubation period for coronavirus disease 2019 (COVID-19) is believed to extend to 14 days, with a median time of 4-5 days from exposure to symptomatic onset. In one study, 97.5% of symptomatic patients developed symptoms within 11.5 days of becoming infected. Most patients with coronavirus disease 2019 (COVID-19) will experience the following (in descending frequency): Fever, Cough, Fatigue, Anorexia, Shortness of breath, Sputum production, Myalgia.

Atypical presentations have been described, and older adults and persons with medical comorbidities may have delayed presentation of fever and respiratory symptoms.

Less common symptoms (< 10%) include headache, confusion, rhinorrhea, sore throat, and hemoptysis. Some patients have experienced gastrointestinal symptoms such as diarrhoea and nausea prior to developing fever and lower respiratory tract signs and symptoms. anosmia may precede the onset of respiratory symptoms. The most common serious manifestation of COVID-19 upon the initial presentation is pneumonia. Fever, cough, dyspnea, and abnormalities on chest imaging are common in these cases. Bilateral distribution of ground-glass opacities (GGO) with or without consolidation in posterior and peripheral lungs was the cardinal hallmark of COVID-19. However, with further analysis of increasing cases, a diversity of interesting CT imaging features were found, including crazy paving pattern, airway changes, halo sign, Pleural changes including pleural thickening and pleural effusion, Vascular enlargement, Air bubble sign, Lymphadenopathy, etc, which may shed light on the possible mechanism of lung injury in COVID-19. On the laboratory aspect leukopenia, leukocytosis, and lymphopenia were common among early cases. Lactate dehydrogenase and ferritin levels are commonly elevated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID 19 PCR positive

Exclusion Criteria:

* Patients less than 18 years of age .

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients diagnosed as COVID19 pneumonia and eligible for search criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | through study completion, an average of 1 year
  Patients assessment using CURB 65|(confusion ,urea level, respiratory rate blood pressure,age above 65 years) score 0 or 1 out patient -2 inpatient observation- 3 or more ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Mokhtar, Study Director — Assiut University; Mostafa kamal, Study Director — Assiut University